CLINICAL TRIAL: NCT01995773
Title: Glucose Metabolism, Adrenal Function, Cortisol Metabolism, Body Composition Physical Activity, and Quality of Life in Healthy Women
Brief Title: Glucose Metabolism and Quality of Life in Healthy Women
Acronym: Healthywomen
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Marianne Andersen, DMSci, Odense University Hospital
Other Study IDs: 280278; 280278 (Other: Odense University Hospital)
Record Dates: First submitted 2013-11-21; First posted 2013-11-27 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2013-11

CONDITIONS: Healthy
Keywords: Healthy women; Quality of life; Glucose metabolism; Adrenal reactivity; Physical activity; Body Composition
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood and urine samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Controls: Healthy control women

SUMMARY:
Polycystic ovary syndrome (PCOS) is a common endocrine disorder in premenopausal women. Women with PCOS often have problems with fertility, unwanted hair growth, and irregular menstrual cycle. PCOS is associated with obesity, changes in glucose metabolism and low quality of life.

In the present study, hormonal profile, glucose metabolism, adrenal functon, androgen levels, cortisol metabolism, anflammatory response, ovarian morphology, body composition, pfysical activity and quality of life is studied in 40 healthy women. The results will be compared with results from studies on women with PCOS in order to investigate any differences in these parametres.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* No medications
* regular menstrual cycle
* no hair growth problems
* BMI 18-35 kg/m2

Exclusion Criteria:

* medication
* diabetes mellitus
* signs of PCOS
* BMI < 18 or > 35

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 40 healthy women with regular menstrual cycle, normal hair growth, and body mass index between 18 and 35 kg/m2
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-12; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Level of androgens | baseline
  Level of testosterone and sexual hormone binding globuline in blood samples

SECONDARY OUTCOMES:
Quality of life | Baseline
  Quality of life measured by validated questionnaires
Body composition | baseline
  Body composition measured by full body DXA-scan with estimates on lean body mass and fat mass
Bone density | baseline
  Bone density measured by DXA scan of hip and wrist
Glucose tolerance | 5 hours
  Glucose tolerance measured by 5 hour oral glucose tolerance test with blood glucose measurements for 5 hours after oral intake of 75 g glucose

OTHER OUTCOMES:
physical activity | one week
  Physical activity measured by accelerometre
adrenal activity | 1 hour
  Adrenal recativity measured by 1 hour ACTH-stimulation test
Ovarian morphology | at baseline
  Ovarian morphology described by vaginal ultrasound with measurements of ovarian volumen and description of phollicles.

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Mumm, MD, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

REFERENCES:
- [Derived] Mumm H, Altinok ML, Henriksen JE, Ravn P, Glintborg D, Andersen M. Prevalence and possible mechanisms of reactive hypoglycemia in polycystic ovary syndrome. Hum Reprod. 2016 May;31(5):1105-12. doi: 10.1093/humrep/dew046. Epub 2016 Mar 23. PMID 27008892